CLINICAL TRIAL: NCT04589468
Title: Phase 1a/b Trial of Exercise as Interception Therapy for Primary High-Risk Cancer
Brief Title: Researching the Effect of Exercise on Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20-378
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer; Stage I Colorectal Cancer; Stage II Colorectal Cancer; Stage III Colorectal Cancer
Keywords: Breast Cancer; Prostate Cancer; Colorectal Cancer; exercise; ctDNA; 20-378; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-Finding/Escalation (Experimental): Fifty (n=50) post-treatment patients with colorectal cancer or breast cancer, deemed high-risk of relapse. The study will use an adaptive continuous reassessment method (CRM) design to assign patients sequentially at trial entry to one of five escalated doses depending on the feasibility / tolerability of exercise therapy evaluated over the total treatment period. The primary objective of this phase 1a trial is to identify the RP2D of exercise therapy for further evaluation in the phase 1b trial.
  Interventions: Other: Exercise
- Dose Expansion (Experimental): An independent cohort of 30 post-treatment patients with colorectal (n=15) or breast (n=15) cancer deemed high-risk of relapse. This cohort expansion trial will only evaluate the RP2D identified in the phase 1a trial. The primary objective of this phase 1b trial is to further evaluate the feasibility, safety, and biological activity of the RP2D.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise therapy in both phases will consist of individualized walking delivered 3 to 6 times weekly (over a 7-day period). Exercise treatment will be delivered for up to 18 months, or until progression of disease or withdrawal of consent, whichever comes first. The phase 1a trial will assess five doses of exercise therapy (i.e., 90, 150, 225, 300, and 375 mins/wk) delivered following a non-linear (i.e., exercise dose is continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period) dosing schedule. The phase 1b trial will only test one dose of exercise therapy - the RP2D identified in the phase 1a trial.

SUMMARY:
Researchers think that exercise may be able to prevent cancer from coming back by lowering ctDNA levels. The purpose of this study is to explore how aerobic exercise (exercise that stimulates and strengthens the heart and lungs and improves the body's use of oxygen) can reduce the level of ctDNA found in the blood. During the study, the highest level of exercise that is practical, is safe, and has positive effects on the body that may prevent the return of cancer (including a decrease in ctDNA levels) will be found. Each level of exercise tested will be a certain number of minutes each week. Once the best level of exercise is found, it will be tested further in a new group of participants. All participants in this study will have been previously treated for breast, prostate, or colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postsurgical diagnosis of patients with primary solid tumors at high-risk of relapse as defined by one of the following:

  ° High-risk primary solid tumor (e.g., colorectal, ovarian, non-small cell lung cancer) (colorectal cancer only for Phase 1a)
* Stage 3 or
* ctDNA positive

  ° High-risk breast cancer
* Residual invasive disease in the breast or the lymph nodes following completion of neoadjuvant chemotherapy (NACT),
* Estrogen receptor (ER), and/or progesterone receptor (PR) positive and HER2 negative,
* CPS-EG score ≥ 3,
* CPS-EG score ≥2 w ith ypN+, or
* Recurrence score ≥ 25
* No evidence of disease
* Age ≥ 18
* Interval of ≥ 1 month but ≤ 2 years following completion of all definitive adjuvant therapy
* Non-exercising (i.e., < 30 minutes of moderate and < 20 mins of vigorous exercise/wk), as assessed by remote activity and heart rate tracking for a 7-day period prior to study entry)

  ° If ≥ 30 minutes but less than 45 minutes of moderate exercise/week, or if ≥ 20 minutes but less than 30 minutes of vigorous exercise/week, patients may be eligible, at the discretion of the PI.
* Cleared for exercise participation as per screening clearance via PAR-Q+
* Willingness to comply with all study-related procedures

Exclusion Criteria:

* Enrollment onto any other interventional investigational study except interventions determined by the PI not to confound study outcomes
* Any other current diagnosis of invasive cancer of any kind
* Distant metastatic malignancy of any kind
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Identify the recommended phase 2 dose (RP2D) of exercise for testing in the phase 1b. | 24 weeks
  Using an adaptive phase 1 (non-randomized) design, non-exercising (i.e., <60 mins/wk of moderate or vigorous exercise) post-treatment patients with primary breast, prostate, or colorectal cancer and detectable ctDNA (n=50) will be administered one of five escalating dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Natera, Inc. (Data or Specimen Analysis Only), San Carlos, California
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04589468/ICF_000.pdf